CLINICAL TRIAL: NCT03880292
Title: SDIM: Spinal Deformity Intraoperative Monitoring. Understanding and Managing Intraoperative Neuromonitoring Changes During Spinal Deformity Surgery: a Prospective Interventional Study
Brief Title: Spinal Deformity Intraoperative Monitoring.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AO Foundation, AO Spine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SDIM
Record Dates: First submitted 2019-03-13; First posted 2019-03-19 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Spinal Deformity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraoperative Maneuvers (Other): To document intraoperative maneuvers performed in repsonse to alerts
  Interventions: Procedure: Document intraoperative Maneuvers

INTERVENTIONS:
Procedure: Document intraoperative Maneuvers — Monitoring procedure during surgery

SUMMARY:
A multicenter, international prospectively collected patient cohort undergoing high-risk spinal cord level surgery or spinal osteotomy procedures will be enrolled to establish the incidence of intraoperative alerts in high-risk spinal cord cases, and explore factors associated with mitigating injury. Baseline, intraoperative, and postoperative characteristics, including demographics, radiological features, lower extremity motor score (LEMS), procedure, anesthetic agents used, and baseline blood pressure will be recorded for either adult patients or pediatric patients.

DETAILED DESCRIPTION:
A multicenter, international prospectively collected patient cohort undergoing high-risk spinal cord level surgery or spinal osteotomy procedures will be enrolled to establish the incidence of intraoperative alerts in high-risk spinal cord cases, and explore factors associated with mitigating injury. Baseline, intraoperative, and postoperative characteristics, including demographics, radiological features, lower extremity motor score (LEMS), procedure, anesthetic agents used, and baseline blood pressure will be recorded for either adult patients or pediatric patients.

If a major change occurs in the intraoperative neuromonitoring, defined as a loss of amplitude greater than 50% in the MEP or SSEP from baseline or sustained EMG activity, a separate form (Appendix 3, Intraoperative Alert Form) will be completed in real-time by the neuromonitoring technician outlining the timing of the alert, blood pressure at the time, surgical events at the time of the change, intraoperative maneuvers performed to address the change, and resultant outcome of these maneuvers to address the neuromonitoring change. For each alert occurring during the procedure, a separate form will be completed.

Once the patient is awake from anesthesia, the treating surgeon will perform a neurological examination to identify details about the deficit including sidedness, LEMS, sensory deficit, injury to the nerve root, incomplete spinal cord (ie anterior cord, posterior cord, central cord, Brown-Sequard), complete spinal cord injury, conus or cauda equina deficit. The examination is repeated on the day of discharge from hospital, or at day 30, whichever comes first and documented in the corresponding form.

The objective of this study is to identify the incidence of intraoperative alerts in high-risk spinal cord cases, correlate significant neuromonitoring changes to intraoperative events, and identify maneuvers that will restore the neuromonitoring changes to baseline. The information provided by this study will educate spinal surgeons to recognize a spinal cord at risk and to perform intraoperative maneuvers that will decrease the incidence of neurological injuries.

ELIGIBILITY:
Inclusion Criteria:

* Age >10 years to <80 years
* Neurologically intact spinal cord (with or without radiculopathy)
* Undergoing primary or revision procedure in the spine
* Anterior and/or posterior surgical approach for any of the following:

  * Correction of spinal deformity with a major Cobb angle of ≥ 80° in the coronal or sagittal plane
  * Correction of high grade spondylolisthesis (Grades 3- 5)
  * Posterior column or 3-column osteotomy
* Requiring multimodal neuromonitoring with EMG, SSEP, and MEP as per standard of care
* Informed consent obtained for patients i.e.:

  * Ability to understand the content of the patient information
  * Willingness and ability to participate in the clinical investigation according to the Clinical Investigation Plan (CIP)
  * Signed and dated EC/IRB approved written informed consent OR
  * Written consent obtained according to defined and IRB/EC approved procedures for patients who are not able to provide independent written informed consent

Exclusion Criteria: • Neurodegenerative disease

* Upper motor neuron lesion
* Growing rods or growth guidance procedures
* Tether or staple procedures
* Stand-alone cervical deformity correction procedures
* Any not medically managed severe systemic disease
* Recent history of substance abuse (ie recreational drugs, alcohol) that would preclude reliable assessment
* Pregnancy or women planning to conceive within the study period
* Prisoner
* Participation in any other medical device or medicinal product study that could influence the results of the present study

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 569 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Number of intraoperative neuromontoring alerts | Intraoperative
  Number of intraoperative neuromonitoring alert, defined as a major change in neuromonitoring signals:
  * SSEP: amplitude loss > 50%
  * MEP: amplitude loss > 50% in two of three muscle groups and/or
  * EMG: sustained activity for > 10 seconds

SECONDARY OUTCOMES:
Intraoperative monitoring alert | Intraoperative
  Intraoperative monitoring alerts:
  • Degree of change in the monitoring signals (SSEP, MEP, EMG)
Success rate of reversal maneuvers to restore signal above the threshold | Intraoperative
  Number and type of maneuver(s) in response to an alert
  * number and type of successful maneuvers
  * number and type of unsuccessful maneuvers
Neurological status | Baseline up to 30 days postoperative
  Neurological status:
  • ASIA Lower extremity motor and sensory score including if a spinal cord syndrome is applicable. A scale from 0 to 5 points in which 0 denotes total paralysis and 5 normal active movement. Sensory will be meassured as either normal, altered or absent.
Timing of intraoperative monitoring alerts | Intraoperative
  Timing: Minutes since skin incision and minutes until recovery in MEP and SSEP

CONTACTS AND LOCATIONS:
Locations (24):
- United States (5):
  - UC San Franciisco, San Francisco, California
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Virginia, Charlottesville, Virginia
- Royal North Shore Hospital, Saint Leonards, Australia
- Brazil (2):
  - Hospital Infantil Joana de Gusmão, Florianópolis
  - Hospital das clinicas de São Paulo e AACD, São Paulo
- Canada (3):
  - Shriners Hospital for Children, Montreal
  - Montreal General Hospital, Montreal
  - Toronto Western Hospital, Toronto
- Nanjing Drum Tower Hospital, Nanjing, China
- Queen Mary Hospital, Hong Kong, Hong Kong
- India (2):
  - Mallika Spine Centre, Guntur
  - Kothari Medical Centre, Kolkata
- Tel Aviv Medical Center - Dana Children's Hospital, Tel Aviv, Israel
- Hamamatsu University School of Medicine, Hamamatsu, Japan
- University Medical Center St. Radboud, Nijmegen, Netherlands
- Ghurki Trust Teaching Hospital, Lahore, Pakistan
- Hospital Vall d'Helbron, Barcelona, Spain
- Acibadem Maslak Hospital, Istanbul, Turkey (Türkiye)
- United Kingdom (3):
  - Guys Hospital, London
  - Salford Royal Hospital, Manchester
  - Nottingham Queens Medical Centre, Nottingham